CLINICAL TRIAL: NCT00673517
Title: The Effect of High Frequency Oscillation on Biological Markers of Ventilator Induced Lung Injury (VILI): Nested Translational Biology Sub-Study of the OSCILLATE Pilot Study
Brief Title: The Effect of High Frequency Oscillation on Biological Markers of Lung Injury
Status: Completed | Type: Observational
Sponsor: Unity Health Toronto (Other)
Collaborators: Canadian Intensive Care Foundation (Other)
Responsible Party: Claudia DosSantos, MD, FRCPC, St. Michael's Hospital
Other Study IDs: OSCILLATE Biomarkers Substudy
Record Dates: First submitted 2008-05-05; First posted 2008-05-07 (Estimated); Last update posted 2008-11-17 (Estimated); Status verified 2008-11

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: Acute respiratory distress syndrome; Ventilator induced lung injury; High frequency oscillation; Lung protective ventilation; Biomarkers; Biotrauma
MeSH Terms: conditions — Respiratory Distress Syndrome; Ventilator-Induced Lung Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Known biomarkers: IL6, IL8, IL10, IL-1Beta, ICAM-1, TGFBeta, Chemokine ligand 10, FGFBeta, VEGF, and INFGamma Novel biomarkers: ACE, surfactant protein D, clara cell protetin, von Willerbrand Facotr, Ang1, Ang2, and TF, PCIII, neuropeptide Y, PBEF, APCRc, and PAI-1
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Patients randomized to high frequency oscillation
- 2: Patients randomized to conventional lung protective ventilation

SUMMARY:
Although mechanical ventilation is life saving, it is associated with a number of severe complications collectively referred to as ventilator induced lung injury (VILI). VILI contributes to the high morbidity and mortality associated with the acute respiratory distress syndrome (ARDS). Within the context of a randomized study evaluating the feasibility of conducting a study comparing high frequency oscillation to conventional lung protective ventilation in early severe ARDS, we are evaluating the effect of both ventilator strategies on biological markers of VILI.

DETAILED DESCRIPTION:
Specific objectives:

To measure known biomarkers conventionally associated with VILI and biotrauma To measure potential novel biomarkers of VILI and biotrauma To identify the best time point for biomarker measurement To collect and store samples for differential expression and genomic analysis

ELIGIBILITY:
Inclusion Criteria:

Informed consent previously obtained for enrollment in the OSCILLATE study:

1. Acute onset of respiratory failure
2. Endotracheal intubation or tracheostomy
3. Hypoxemia (P:F <200 mmHg)
4. Bilateral alveolar consolidation

Exclusion Criteria:

1. Refusal of consent to participate in this biomarkers substudy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subset of patients enrolled in the parent study (OSCILLATE- #NCT00474656) Patients enrolled in the parent study have early severe acute respiratory syndrome and will be recruited from a critical care environment
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2007-11; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Serum concentration of known biomarkers associated with VILI and biotrauma | Baseline, after standardization, 6-10 hours after randomization, 12-16 hours after randomization, 24-30 hours after randomization, 72-76 hours after randomization, and every 3 subsequent days until death, discharge, or completion of the study at 28 days

SECONDARY OUTCOMES:
Serum concentration of tissue and cell specific markers that are potential novel biomarkers associated with VILI and biotrauma | Baseline, after standardization, 6-10 hours after randomization, 12-16 hours after randomization, 24-30 hours after randomization, 72-76 hours after randomization, and every 3 subsequent days until death, discharge, or completion of the study at 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Claudia C DosSantos, MD, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada